CLINICAL TRIAL: NCT01927939
Title: The Effectiveness of 18F-FDG PET Metabolic Phenotype in Evaluating Therapeutic Response for Breast Cancer Patients With Bone Metastases.
Brief Title: 18F-FDG PET Metabolic Phenotype in Evaluating Therapeutic Response for Breast Cancer Patients With Bone Metastases.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201207002MIB
Record Dates: First submitted 2013-08-16; First posted 2013-08-23 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer; 18F-FDG PET
Keywords: Breast cancer; bone metastases; 18F-FDG PET; 99mTc bone scintigraphy; therapy response monitoring; prognosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Histological proven breast cancer with bone lesion

SUMMARY:
This study is to evaluate the effectiveness of 18F-FDG PET in following up of metastastic bone lesions and in predicting outcome for breast cancer patients after therapy.

Primary outcome: Using 18F-FDG uptake to evaluate the metastatic bone status after treatment. The PET results will be compared with the results in Tc-99m MDP bone scintigraphy.

Secondary outcome: Evaluate the relationship between the 18F-FDG uptake of the metastatic bone lesions and (1) breast cancer related tumor marker, (2) patients' survival.

DETAILED DESCRIPTION:
Background: Although 99mTc MDP bone scintigraphy is a sensitive tool for screening metastatic bone status, it is not a satisfactory imaging modality in evaluating residual disease after therapy. 18F-FDG PET has been an effective imaging tool for many malignancies including breast cancer, not only in diagnosis and staging, but also in monitoring response and following up disease status after therapy.

Purpose: This study is to evaluate the effectiveness of 18F-FDG PET in following up of metastastic bone lesions and in predicting outcome for breast cancer patients after therapy.

Method: Breast cancer patients with bone metastases, age 20-90 year-old, will be included in this study.

Primary outcome: Using 18F-FDG uptake to evaluate the metastatic bone status after treatment. The PET results will be compared with the results in Tc-99m MDP bone scintigraphy.

Secondary outcome: Evaluate the relationship between the 18F-FDG uptake of the metastatic bone lesions and (1) breast cancer related tumor marker, (2) patients' survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age：20-90 years old
2. Histological proven breast cancer, with known metastatic bone lesion(s)
3. written informed consent signed

Exclusion Criteria:

1. pregnant or intend to be pregnant
2. other malignancies known

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histological proven breast cancer, with known metastatic bone lesion(s)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The uptake of 18F-FDG PET. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yen Ruoh Fang, M.D.,Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Solomayer EF, Diel IJ, Meyberg GC, Gollan C, Bastert G. Metastatic breast cancer: clinical course, prognosis and therapy related to the first site of metastasis. Breast Cancer Res Treat. 2000 Feb;59(3):271-8. doi: 10.1023/a:1006308619659. PMID 10832597
- [Background] Roberts CC, Daffner RH, Weissman BN, Bancroft L, Bennett DL, Blebea JS, Bruno MA, Fries IB, Germano IM, Holly L, Jacobson JA, Luchs JS, Morrison WB, Olson JJ, Payne WK, Resnik CS, Schweitzer ME, Seeger LL, Taljanovic M, Wise JN, Lutz ST. ACR appropriateness criteria on metastatic bone disease. J Am Coll Radiol. 2010 Jun;7(6):400-9. doi: 10.1016/j.jacr.2010.02.015. PMID 20522392
- [Background] Houssami N, Costelloe CM. Imaging bone metastases in breast cancer: evidence on comparative test accuracy. Ann Oncol. 2012 Apr;23(4):834-43. doi: 10.1093/annonc/mdr397. Epub 2011 Sep 6. PMID 21896542
- [Background] Vassiliou V, Andreopoulos D, Frangos S, Tselis N, Giannopoulou E, Lutz S. Bone metastases: assessment of therapeutic response through radiological and nuclear medicine imaging modalities. Clin Oncol (R Coll Radiol). 2011 Nov;23(9):632-45. doi: 10.1016/j.clon.2011.03.010. Epub 2011 Apr 29. PMID 21530193
- [Background] Galasko CS. Diagnosis of skeletal metastases and assessment of response to treatment. Clin Orthop Relat Res. 1995 Mar;(312):64-75. PMID 7634619
- [Background] Cook GJ, Fogelman I. The role of nuclear medicine in monitoring treatment in skeletal malignancy. Semin Nucl Med. 2001 Jul;31(3):206-11. doi: 10.1053/snuc.2001.23527. PMID 11430527
- [Background] Vogel CL, Schoenfelder J, Shemano I, Hayes DF, Gams RA. Worsening bone scan in the evaluation of antitumor response during hormonal therapy of breast cancer. J Clin Oncol. 1995 May;13(5):1123-8. doi: 10.1200/JCO.1995.13.5.1123. PMID 7537797
- [Background] Rossleigh MA, Lovegrove FT, Reynolds PM, Byrne MJ, Whitney BP. The assessment of response to therapy of bone metastases in breast cancer. Aust N Z J Med. 1984 Feb;14(1):19-22. doi: 10.1111/j.1445-5994.1984.tb03578.x. PMID 6235799
- [Background] Mitsudomi T, Kosaka T, Endoh H, Horio Y, Hida T, Mori S, Hatooka S, Shinoda M, Takahashi T, Yatabe Y. Mutations of the epidermal growth factor receptor gene predict prolonged survival after gefitinib treatment in patients with non-small-cell lung cancer with postoperative recurrence. J Clin Oncol. 2005 Apr 10;23(11):2513-20. doi: 10.1200/JCO.2005.00.992. Epub 2005 Feb 28. PMID 15738541
- [Background] Tateishi U, Gamez C, Dawood S, Yeung HW, Cristofanilli M, Macapinlac HA. Bone metastases in patients with metastatic breast cancer: morphologic and metabolic monitoring of response to systemic therapy with integrated PET/CT. Radiology. 2008 Apr;247(1):189-96. doi: 10.1148/radiol.2471070567. PMID 18372468
- [Background] Du Y, Cullum I, Illidge TM, Ell PJ. Fusion of metabolic function and morphology: sequential [18F]fluorodeoxyglucose positron-emission tomography/computed tomography studies yield new insights into the natural history of bone metastases in breast cancer. J Clin Oncol. 2007 Aug 10;25(23):3440-7. doi: 10.1200/JCO.2007.11.2854. Epub 2007 Jun 25. PMID 17592153
- [Background] Israel O, Goldberg A, Nachtigal A, Militianu D, Bar-Shalom R, Keidar Z, Fogelman I. FDG-PET and CT patterns of bone metastases and their relationship to previously administered anti-cancer therapy. Eur J Nucl Med Mol Imaging. 2006 Nov;33(11):1280-4. doi: 10.1007/s00259-006-0141-3. Epub 2006 Jun 22. PMID 16791597
- [Background] De Giorgi U, Mego M, Rohren EM, Liu P, Handy BC, Reuben JM, Macapinlac HA, Hortobagyi GN, Cristofanilli M, Ueno NT. 18F-FDG PET/CT findings and circulating tumor cell counts in the monitoring of systemic therapies for bone metastases from breast cancer. J Nucl Med. 2010 Aug;51(8):1213-8. doi: 10.2967/jnumed.110.076455. Epub 2010 Jul 21. PMID 20660382